CLINICAL TRIAL: NCT02160457
Title: Instrumented Gait Analysis and Individually Tailored Interdisciplinary Interventions for Children With Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Gait Analysis and Interdisciplinary Interventions for Children With Cerebral Palsy
Acronym: CPinMotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Sonderborg Hospital (Other Government); Sygehus Lillebaelt (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); University of Salford (Other); Region of Southern Denmark (Other); Ludvig and Sara Elsass Foundation (Unknown); Association of Danish Physiotherapists (Other)
Responsible Party: Principal Investigator, Helle Mätzke Rasmussen, Ph.d. Student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20120162
Record Dates: First submitted 2014-06-02; First posted 2014-06-10 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Instrumented gait analysis; Gait Deviation Index
MeSH Terms: conditions — Cerebral Palsy | interventions — Methods; Immunoglobulin A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention with IGA (Experimental): Individually tailored interdisciplinary intervention based on measures performed as part of the Cerebral Palsy follow-Up Program and other clinical examinations AND instrumented gait analysis (IGA)
  Interventions: Other: Intervention with IGA
- Intervention without IGA (No Intervention): 'Care as usual' - Individually tailored interdisciplinary interventions based on measures performed as part of the Cerebral Palsy follow-Up Program and other clinical examinations BUT NOT (IGA).

INTERVENTIONS:
Other: Intervention with IGA — Individually tailored interdisciplinary intervention based on measures performed as part of the Cerebral Palsy follow-Up Program and other clinical examinations AND instrumented gait analysis
  The instrumented gait analysis consists of four steps:
  1. Instrumented gait analysis (data collection with a 8-camera Vicon T40 system (Vicon, Oxford, UK) and 2 force plates (AMTI, OR6-7-1000)
  2. Impairment-Focused Interpretation
  3. Recommendation for interdisciplinary interventions
  4. Dissemination of recommendations
  The two modalities differs in the use of IGA, but the study is not indented to document the effect of IGA alone, but to document the difference in the effects of the interdisciplinary interventions, when IGA is implemented to the experimental group.
  Other Names: Vicon T40 system, Vicon, Oxford, UK; Advanced Mechanical Technology Inc. (AMTI), OR6-7-1000, Watertown, USA
  Arms: Intervention with IGA

SUMMARY:
The aim of this study is to test the hypothesis, that improvements in gait pattern following individually tailored interventions guided by instrumented 3-dimensional gait analysis are superior to those used in 'care as usual'.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) who walk independently often have an altered gait pattern. Interdisciplinary interventions in terms of orthopaedic surgery, spasticity management, physical therapy and orthotics aim to improve the gait pattern. Standardised measurements are used in the Cerebral Palsy follow-Up Program to assess walking. However, these measurements do not describe features in the gait pattern reflecting underlying neuro-musculoskeletal impairments. This can be done with instrumented 3-dimensional gait analysis (IGA). It has never been investigated whether interdisciplinary interventions designed to address impairments identified by IGA result in improved gait pattern compared with 'care as usual' without IGA in children with CP. The aim of this study is to test the hypothesis, that improvements in gait pattern following individually tailored interventions guided by IGA are superior to those used in 'care as usual'.

A prospective, single blind, randomised, parallel group study will be conducted. Participants will be recruited from the Cerebral Palsy follow-Up Program. Children aged 5 to 9 years with spastic CP, classified at Gross Motor Function Classification System levels I or II will be included. The interventions under investigation are 1) Individually tailored interdisciplinary intervention addressing impairments identified by IGA and 2) 'care as usual' (interdisciplinary interventions without IGA). The primary outcome is gait pattern measured by the Gait Deviation Index. Secondary outcome measures are, walking performance and patient-reported outcomes of functional mobility, health-related quality of life and overall health, pain and participation. Explorative outcome measures include walking performance, gait pattern, behavior of health care providers and the applied interventions. The primary endpoint for assessing the outcome of the two interventions will be 52 weeks after start of intervention. A follow up will also be performed at 26 weeks after start of intervention; however, exclusively for the patient-reported outcomes.

To our knowledge, this is the first randomised controlled trial comparing the effects of an individually tailored interdisciplinary intervention designed to address impairments identified by IGA versus 'care as usual' in children with CP. Consequently, the study will provide novel evidence for the use of IGA in interdisciplinary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Spastic Cerebral palsy
* Gross Motor Function Classification System levels I or II.

Exclusion Criteria:

* Earlier interventions in the form of orthopaedic surgery within the past 52 weeks, injection with botulinum toxin type A in the 12 weeks prior to baseline assessments
* Relocation to another region during the trial.
* If the child not are able to demonstrate sufficient co-operation and cognitive understanding to participate in the IGA.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Gait Deviation Index | Baseline, 52 weeks
  Gait Deviation Index (GDI) is based upon kinematic data from the Instrumented Gait Analysis, and is an quantitative index that summarises the overall gait pattern into a single score for each patient by comparison with non-pathological gait. A GDI value of 100 represents the absence of gait pathology, and each 10-point decrement below 100 indicates one standard deviation from normal gait kinematics. For the primary outcome measure, the median of five trials for each leg will be used to calculate the average of both legs to provide a single index for each child.

SECONDARY OUTCOMES:
Change from baseline in 1-minute walk test | Baseline, 52 weeks
  Walking performance is assessed with the 1-minute walk test. The test measure the distance in meters, when the child walks as fast as possible.
Change from baseline in Mobility Scale of the Pediatric Evaluation of Disability Inventory | Baseline, 52 weeks
  The Mobility Scale of the Pediatric Evaluation of Disability Inventory evaluates the child's functional mobility in everyday activities with regard to functional skills and caregiver assistance. The Paediatric Evaluation of Disability Inventory will be applied as a parental questionnaire, allowing comparison of the child's functional skills over time for each of the two dimensions.
Change from baseline in Pediatric Quality of Life Inventory Cerebral Palsy Module | Baseline, 52 weeks
  The Pediatric Quality of Life Inventory Cerebral Palsy Module is a measure of health-related quality of life, specifically designed for children with CP. The Pediatric Quality of Life Inventory Cerebral Palsy Module is based upon the parents' report and measures physical, emotional, social and school functioning.
Change from baseline in Pediatric Outcome Data Collection Instrument | Baseline, 52 weeks
  The Pediatric Outcome Data Collection Instrument assesses overall health, pain and participation in normal daily activities.
Change from baseline in Mobility Scale of the Pediatric Evaluation of Disability Inventory | Baseline, 26 weeks
  The Mobility Scale of the Pediatric Evaluation of Disability Inventory evaluates the child's functional mobility in everyday activities with regard to functional skills and caregiver assistance. The Paediatric Evaluation of Disability Inventory will be applied as a parental questionnaire, allowing comparison of the child's functional skills over time for each of the two dimensions.
Change from baseline in Pediatric Quality of Life Inventory Cerebral Palsy Module | Baseline, 26 weeks
  The Pediatric Quality of Life Inventory Cerebral Palsy Module is a measure of health-related quality of life, specifically designed for children with CP. The Pediatric Quality of Life Inventory Cerebral Palsy Module is based upon the parents' report and measures physical, emotional, social and school functioning.
Change from baseline in Pediatric Outcome Data Collection Instrument | Baseline, 26 weeks
  The Pediatric Outcome Data Collection Instrument assesses overall health, pain and participation in normal daily activities.

OTHER OUTCOMES:
Change from baseline in Gait Variable Score | Baseline, 52 weeks
  The Gait Variable Score is used to measure changes in gait pattern. Gait Variable Score is an index for a single gait variable. The Gait Variable Scores are determined for the following nine variables: Pelvic tilt, pelvic obliquity, pelvic rotation, hip flexion, hip adduction, hip rotation, knee flexion, dorsiflexion and foot progression
Change from baseline in Measure of Processes of Care | Baseline, 52 weeks
  Measure of Processes of Care is a self-report measure of parents' perception of the extent to which the health services that their child receives are family-centred.
Applied interventions | 52 weeks
  Records from the Cerebral Palsy Follow-Up Program of the applied interventions will be used to explore differences (used vs. not used) in the use of the following intervention categories in the two groups: Orthopaedic surgery, Spasticity management, Physical Therapy and Orthotics.
Difference in recommended and applied interventions | Baseline, 52 weeks
  Records from the Cerebral Palsy Follow-Up Program of the recommended and actually applied interventions in the experimental group will be used to explore the differences (used vs. not used) in the recommended and actually applied interventions in regard to the following categories: Orthopaedic surgery, Spasticity management, Physical Therapy and Orthotics.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Rasmussen, Ph.d. stud., Principal Investigator — University of Southern Denmark and Odense University Hospital; Anders Holsgaard-Larsen, Ph.d., Study Chair — University of Southern Denmark and Odense University Hospital
Locations (1):
- University of Southern Denmark - Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Fonvig CE, Rasmussen HM, Overgaard S, Holsgaard-Larsen A. Effectiveness of instrumented gait analysis in interdisciplinary interventions on parents' perception of family-centered service and on gross motor function in children with cerebral palsy: a randomized controlled trial. BMC Pediatr. 2020 Sep 1;20(1):411. doi: 10.1186/s12887-020-02315-2. PMID 32873289
- [Derived] Rasmussen HM, Pedersen NW, Overgaard S, Hansen LK, Dunkhase-Heinl U, Petkov Y, Engell V, Baker R, Holsgaard-Larsen A. The use of instrumented gait analysis for individually tailored interdisciplinary interventions in children with cerebral palsy: a randomised controlled trial protocol. BMC Pediatr. 2015 Dec 7;15:202. doi: 10.1186/s12887-015-0520-7. PMID 26643822

DOCUMENTS (2):
  • Statistical Analysis Plan: Primary analysis (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT02160457/SAP_000.pdf
  • Statistical Analysis Plan: Secondary analysis on tertiary outcome measures (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02160457/SAP_001.pdf